CLINICAL TRIAL: NCT03891550
Title: Micro-elimination of Hepatitis C Virus Infection With Pan-genotypic DAA Regimen in Hepatitis C Highly Endemic and Contagious Community (ERASE-C)
Brief Title: Micro-elimination of Hepatitis C Virus Infection in Uremics
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20180057
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis C
Keywords: HCV, micro-elimination, DAA
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Intervention Model Description: active, open labeled, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOF/VEL (Experimental): sofosbuvir (SOF) 400 mg/Velpatasvir(VEL) 100 mg fixed-dosage combination once-daily for 12 weeks
  Interventions: Drug: Epclusa

INTERVENTIONS:
Drug: Epclusa — sofosbuvir (SOF) 400 mg/Velpatasvir(VEL) 100 mg fixed-dosage combination once-daily for 12 weeks for all HCV genotype patients with and without hepatic decompensation

SUMMARY:
There is a huge gap between the clinical efficacy and community effectiveness in the treatment of chronic hepatitis C in Taiwan. HCV infection prevails in uremic patients with the prevalence of > 10 % in Taiwan.The current study will be executed in each participating hemodialysis centers by an outreach team of HCV treaters, treating all of the HCV-viremic uremia patients and HD staffs at the same time (group therapy) in each individual HD center (Erase-C campaign) with all oral directly-acting antivirals, to ensure the rates of diagnosis, accessibility, treatment and follow-up.The purpose of the study is to demonstrate a model of care using outreach HCV treaters by implementing the concept of "group therapy" with one-size-fit-all pangenotypic DAA regimen, 12 weeks of sofosbuvir/velpatasvir, in each individual hemodialysis center (Erase-C campaign) to achieve HCV micro-elimination.

DETAILED DESCRIPTION:
Background 1.1 Background of ESRD patients on maintenance HD with chronic HCV infection Taiwan has the leading prevalence and incidence of end-stage renal disease (ESRD) worldwide. Uremic patients on maintenance hemodialysis (HD) are at great risk for hepatitis C virus (HCV) infection. The prevalence and annual incidence of HCV infection in ESRD patients undergoing hemodialysis have been reported to be 10%-59% and 0.2%-6.2%, respectively. HCV-related morbidities and mortality remain the major disease burdens in the ESRD population. Uremic patients with HCV infection are associated with higher risk of morbidities and mortality. Anti-HCV therapy at individual patient level might prevent the liver-related morbidity/mortality, however, patients remain at high risk of HCV new- or re-infection if there are HCV patients untreated or failed treatment in the HD units. FORMOSA-LIKE is a study group of Hepatologists and Nephrologists from 15 HD centers at community, regional or tertiary hospitals (now 19) that caring > 1900 uremic patients under maintenance HD in Taiwan, established in 2012. The anti-HCV seropositivity rate was 17% among HD patients; HCV viremic rate was 74.6% among anti-HCV seropositivity HD subjects. To decrease the rate of new HCV infection between HD patients, all anti-HCV-seropositive uremic patients are requested to receive HD in an isolated "HCV-zone". Recently, the Taiwan Center for Disease Control recommends that anti-HCV-seropositive uremic patients could be moved from HCV-zone to clean-zone if they have PCR-undetectable HCV RNA for more than 24 weeks, whatever spontaneously or after antiviral therapy. The new policy raises the question that whether it is possible to create a "NoC-HD" environment where HCV-zone no longer exists due to all HCV-viremic patients are cured. The achievement of NoC-HD could provide not only obligation of transmitting HCV within HD centers, but also a much more cost-effective care of hemodialysis.

1.2 Gap of anti-HCV therapy for HCV patients on maintenance HD There is a huge gap between the clinical efficacy and community effectiveness in the treatment of chronic hepatitis C in Taiwan, with treatment uptake rate < 20%. The treatment hurdle is more significant in uremic patients because many primary HD units outside medical centers have poor accessibility to HCV testing and treatment. Meanwhile, directly acting antivirals (DAAs) has just replaced interferon (IFN)-based therapy as standard of care in Taiwan since 2017. The majority of HD patients do not receive IFN-based therapy due to unsatisfactory efficacy and frequent and significant adverse events. The innovation of DAAs provide very high sustained virological response (SVR) rates of > 95% in general population and uremic patients with chronic HCV infection. Nevertheless, there remains big hurdle for uremic HCV patients to access DAA therapy because that only gastroenterologists specialists could prescribe reimbursed DAA regimens in Taiwan. Sofosbuvir/Velpatasvir (SOF/VEL) is a fixed-dose combination of HCV non-structural 5A (NS5A) inhibitor and NS5B inhibitor. SOF/VEL is the only all oral, pan-genotypic DAA not only for patients with compensated liver disease but also for patients in the decompensated status. A universal 12-week regimen of SOF/VEL provides a SVR12 rate of > 95 % in general population with different viral genotypes and special populations, and is the current standard of care by regional guidelines. SOF/VEL has been recently proved to be highly effective and well tolerated in uremic patients with HCV viremia; an SVR12 rate of 95% could be achieved in uremic patients receiving 12 weeks of SOF/VEL.

1.3 Background of HCV elimination World Health Organization (WHO) sets a goal of HCV elimination worldwide by 2030. However, there remains many barriers to achieve the goal of HCV elimination, including the low rates of disease diagnosis/awareness, accessibility and treatment. The concept of micro-elimination of HCV by using pangenotypic DAA for HCV communities could provide evidence to obviate the treatment barriers to HCV elimination. In addition, the reported annual incidence of new HCV infection among uremic patients under maintenance hemodialysis in Taiwan was 1.36%. Therefore, treatment as prevention; increasing the treatment uptake at the population level would provide completely blockage of HCV spreading in highly endemic/contagious community. The target population of micro-elimination should possess three major characteristics: 1. high prevalence 2. highly contagious 3. closely contact environment. The current uremic population in Taiwan fulfills all the factors mentioned above.

The current study will be executed in each participating hemodialysis centers by an outreach team of HCV treaters, treating all of the HCV-viremic uremia patients and HD staffs at the same time (group therapy) in each individual HD center (Erase-C campaign), to ensure the rates of diagnosis, accessibility, treatment and follow-up.

Objectives:

The purpose of the study is to demonstrate a model of care using outreach HCV treaters by implementing the concept of "group therapy" with one-size-fit-all pangenotypic DAA regimen, 12 weeks of SOF/VEL, in each individual hemodialysis center (Erase-C campaign) to achieve HCV micro-elimination.

Study schedule:

One arm: sofosbuvir (SOF) 400 mg/Velpatasvir(VEL) 100 mg fixed-dosage combination once-daily for 12 weeks for all HCV genotype patients with and without hepatic decompensation HCV RNA and liver function tests, pregnancy test will be monitoring at baseline, during and after treatment

ELIGIBILITY:
Inclusion Criteria:

* Medical staffs and patients on HD, with age 20 years or more at the time of screening, agree to participate the study and provide informed consent.
* A negative serum pregnancy test is required for female subjects (unless permanently sterile or greater than two years post-menopausal)
* Subjects and their partners are considered childbearing potential must agree to use acceptable contraceptive method during treatment till SVR12.
* Ability to participate and willingness to give written informed consent and to comply with the study restrictions.

Exclusion Criteria:

Medical staffs or uremic patients who are seropositive for HCV RNA and have contraindication to or unwilling to receive SOF/VEL, or who failed to prior IFN-free direct antiviral agents (DAA) regimens

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
The rate of HCV micro-elimination in the per-protocol (PP) HD centers | 9 months
  proportion of HD centers t-C campaign"hat achieve an 80% reduction of prevalence rate of HCV viremia in each individual HD center at post campaign week 24 among the HD centers that having ≥ 90% of HCV viremic patients participating the "Erase

SECONDARY OUTCOMES:
Rate of HCV micro-elimination in the full-analysis-set (FAS) HD centers | 9 months
  proportion of HD centers that achieve an 80% reduction of prevalence rate of HCV viremia in each individual HD center at post campaign week 24 among the HD centers that having ≥ one HCV viremic patients participating the "Erase-C campaign" and receiving ≥ one doe of any study medication.
Rate of NoC-HD in the per-protocol (PP) HD centers | 9 months
  proportion of HD centers with all patients of HCV viremia at baseline becoming HCV-RNA < LLOQ, at post campaign week 24 in HD centers that having all HCV viremic patients participating the "Erase-C campaign".
Rate of NoC-HD in the full-analysis-set (FAS) HD centers | 9 months
  proportion of HD centers with all patients of HCV viremia at baseline becoming HCV-RNA < LLOQ, at post campaign week 24 in HD centers that having ≥ one HCV viremic patients participating the "Erase-C campaign" and receiving ≥ one doe of any study medication.
Proportion of drug related adverse events | 6 months
  any adverse events, serious adverse events, discontinuations and laboratory abnormality during and 24 weeks after study medication in the full-analysis-set (FAS) population (subjects receiving ≥ 1 dose of any study medication).
SVR12 rate in the FAS population | 6 months
  proportion of patients with HCV-RNA < LLOQ, at post treatment week 12 in FAS population
SVR rate in the modified full-analysis-set (mFAS) population | 6 months
  proportion of patients with HCV-RNA < LLOQ at posttreatment week 12 in mFAS population (subjects receiving ≥1 dose of any study medication and HCV RNA data available at posttreatment week 12 and excluding non-virological failures)
The annual incidence rate of new HCV infection | 60 months
  new infection of HCV among staffs/patients who are HCV non-viremic at pre-screening of the study, or reinfection characterized by viral sequencing, among HCV staffs/patients who achieve an SVR12 after SOF/VEL treatment, during 5-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, MD.,PhD., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Huang CF, Dai CY, Wang CW, Liang PC, Wei YJ, Tsai PC, Jang TY, Hsu PY, Jia-Jung Lee, Niu SW, Huang JC, Yeh ML, Huang CI, Hsieh MY, Lin YH, Chen SC, Chiu YW, Huang JF, Chang JM, Hwang SJ, Chuang WL, Yu ML; FORMOSA-LIKE investigators. Therapy as prevention toward HCV elimination in maintenance hemodialysis: a multi-center, prospective cohort study. Clin Kidney J. 2023 Jun 14;16(12):2429-2436. doi: 10.1093/ckj/sfad138. eCollection 2023 Dec. PMID 38046041
- [Derived] Yu ML, Huang CF, Wei YJ, Lin WY, Lin YH, Hsu PY, Hsu CT, Liu TW, Lee JJ, Niu SW, Huang JC, Hung TS, Yeh ML, Huang CI, Liang PC, Hsieh MY, Chen SC, Huang JF, Chang JM, Chiu YW, Dai CY, Hwang SJ, Chuang WL; FORMOSA-LIKE investigators. Establishment of an outreach, grouping healthcare system to achieve microelimination of HCV for uremic patients in haemodialysis centres (ERASE-C). Gut. 2021 Dec;70(12):2349-2358. doi: 10.1136/gutjnl-2020-323277. Epub 2020 Dec 10. PMID 33303567